CLINICAL TRIAL: NCT07260162
Title: A First In Human Phase I Trial Evaluating Safety, Tolerability and Response of [211At]At-Girentuximab (ATO-101™) in Patients With Non-Muscle-Invasive Bladder Cancer Refractory to Standard Treatment
Brief Title: Evaluation of Safety, Tolerability and Response of ATO-101™ in Patients With Non-Muscle-Invasive Bladder Cancer (PERSEVERANCE EU)
Acronym: PERSEVERANCE
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICO-2023-18
Record Dates: First submitted 2025-11-19; First posted 2025-12-03 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Bladder Cancer
Keywords: Non-Muscle-Invasive Bladder cancer (NMIBC); Girentuximab; Astatine 211; Phase I; First In Human (FIH); Carbonic anhydrase IX (CAIX); Intravesical instillation; [211At]At-Girentuximab; ATO-101™
MeSH Terms: conditions — Urinary Bladder Neoplasms; Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Intervention Model Description: ATO-101™ is an anti-CA-IX antibody (Girentuximab) radiolabeled with an alpha-emitting radionuclides (astatine-211)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ATO-101™ (Experimental): [211At]At-Girentuximab (ATO-101™) intravesical administration
  Interventions: Drug: ATO-101™

INTERVENTIONS:
Drug: ATO-101™ — The study drug: [211At]At-Girentuximab (ATO-101™) is administered via intravesical instillation
  Other Names: [211At]At-Girentuximab

SUMMARY:
Non-Muscle-Invasive Bladder cancer (NMIBC) tumours often recur despite TransUrethral Resection of Bladder (TURB) and Bacillus Calmette-Guerin (BCG) intravesical instillations, and have no effective conservative treatment options. Alpha emitters like Astatine-211 (211At), due to their short path and short half-life, show promise for superficial targets such as NMIBC.

Carbonic anhydrase IX (CAIX), overexpressed in 70-90% of NMIBC cases but absent in healthy tissues, is an ideal target.

A clinical feasibility Positron emission tomography-computed tomography (PET/CT) imaging study (Pertinence, NCT04897763) was conducted at Institut de cancérologie Ouest (ICO) in six patients using Girentuximab labelled with Zirconium-89 ([89Zr]Zr-girentuximab). It demonstrated successful tracer targeting and no radioactive leakage beyond the bladder following intravesical instillation. The study also confirmed the absence of toxicity, contamination, or significant additional staff radiation exposure.

ATO-101™ ([²¹¹At]At-girentuximab) could enable localised tumour destruction while preserving the bladder in patients with BCG-unresponsive NMIBC. The ongoing First In Human (FIH) study evaluate the safety of ATO-101™ in patients with BCG-unresponsive NMIBC.

ELIGIBILITY:
Inclusion Criteria:

* Performance Status (PS): 0 or 1.
* Patient experiencing relapse following standard treatment (BCG therapy with or without Mitomycin), before radical surgery which is being considered as a therapeutic option.
* Clinical evidence of NMIBC based on cystoscopy and proven histologically of papillary tumours.
* Histologically confirmed bladder cancer patients relapsing without muscle invasion.
* Negative serum/urine pregnancy test prior to ATO-101™ administration for female patient of childbearing potential.
* Consent to use a contraception method for at least 3 months after administration of ATO-101™.
* Adequate organ function confirmed by laboratory tests results allowing for safe administration of ATO-101™.

Exclusion Criteria:

* Patient with urinary incontinence.
* Patient treated with anticoagulant or platelet antiaggregant therapies.
* Symptoms of urine infection.
* Patient with urethral stenosis.
* Patient with valvular heart disease.
* No history of congestive heart failure.
* Known hypersensitivity to Girentuximab.
* Exposure to any experimental diagnostic or therapeutic drug within 30 days prior the date of planned administration of ATO-101™.
* Serious non-malignant disease that may interfere with the objectives of the study or with the safety or compliance of the patient as judged by the investigator.
* Concomitant cancer in the past 5 years except cutaneous cancers (except melanoma) and in situ carcinoma in past 3 years.
* Prior chemotherapy, radiotherapy (other than short cycle of palliative radiotherapy), immunotherapy within 21 days of ATO-101™ administration.
* Pregnant or likely to be pregnant or nursing patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
To determine the Maximum Tolerated Dose (MTD) of ATO-101™. | 15 days
  The primary endpoint is the occurrence of dose-limiting toxicities (DLTs) during the DLT observation period.
To determine the Recommended Dose for Expansion (RDE) of ATO-101™. | 15 days
  The primary endpoint is the occurrence of dose-limiting toxicities (DLTs) during the DLT observation period.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline ROUSSEAU, MD, PhD, Principal Investigator — Institut de Cancérologie de l'OUEST _ ICO
Locations (1):
- Institut de Cancérologie de l'Ouest, Saint-Herblain, Loire Atlantique, France